CLINICAL TRIAL: NCT02812888
Title: Serum Betatrophin Levels and Its Influencing Factors in Patients With Hyperthyroidism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hu Hao (Other)
Responsible Party: Sponsor-Investigator, Hu Hao, Deputy Director, Department of endocrinology, Principal Investigator, Clinical Associate Professor, The First People's Hospital of Xuzhou
Organization: The First People's Hospital of Xuzhou (Other)
Other Study IDs: FirstPHXuzhou; ChiCTR (Registry Identifier: 16008506)
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Hyperthyroidism
Keywords: Hyperthyroidism; Betatrophin
MeSH Terms: conditions — Hyperthyroidism | interventions — Methimazole; Propylthiouracil; Propranolol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hyperthyroid Patients: Patients with hyperthyroidism
  Interventions: Drug: thionamide treatment for 3 months
- NC group: Normal control subjects

INTERVENTIONS:
Drug: thionamide treatment for 3 months — Hyperthyroid patients would received thionamide treatment (methimazole, propylthiouracil, or propranolol) for 3 months, and euthyroidism would be obtained.
  Other Names: methimazole, propylthiouracil, or propranolol
  Groups: Hyperthyroid Patients

SUMMARY:
Clustering of various metabolic parameters including abdominal obesity, hyperglycaemia, low high-density lipoprotein cholesterol, elevated triglycerides and hypertension have been used worldwide as metabolic syndrome to predict cardiometabolic risk. Thyroid dysfunction impacts on various levels of these components.

Recent evidence from HepG2 cells indicates that betatrophin, also known as TD26/RIFL/lipasin/ANGPTL8/C19orf80, a secreted protein that regulates glucose, lipid metabolism, and energy homeostasis, is induced by T3. However, the role of betatrophin in hyperthyroid patients is unknown.

The objective was to study serum betatrophin levels in hyperthyroid patients and the association of serum betatrophin levels with hyperthyroidism.

DETAILED DESCRIPTION:
Thyroid hormone (TH) is a critical hormone responsible for growth, development, and metabolism. It maintains basal metabolic rate (BMR), improves adaptive thermogenesis, and thus modulates body weight by fine-tuning energy expenditure and intake. Hyperthyroidism, a condition with excess TH, presents a status of negative energy balance that is characterized by weight loss, increased energy expenditure, and accelerated lipolysis and gluconeogenesis. The mechanism underlying hypermetabolic status in hyperthyroidism is complicated. In hyperthyroidism, excess TH promotes the metabolism rate primarily by binding to TH receptor α or β, and in turn by further influencing diverse metabolic pathways. Recent studies have revealed that TH signals were involved in cross talk with a range of other metabolic signaling pathways in different metabolic organs. In liver, TH interacts with peroxisome proliferator-activated receptor (PPAR) α, PPARγ, and liver X receptor α pathway; promotes fatty acid oxidation; decreases cholesterol; and enhances gluconeogenesis. The elements required for TH action are well documented, but understanding the interaction between TH and various pathways remains a challenge.

Betatrophin, also known as TD26/RIFL/lipasin/ANGPTL8/C19orf80, is a novel protein predominantly expressed in human liver. Increasing evidence has revealed associations between betatrophin expression, glycemia and serum lipid profiles, particularly in patients with obesity or diabetes. Stimulators of betatrophin, such as insulin, thyroid hormone, irisin, SIRT1 and caloric intake, are usually relevant to energy expenditure or thermogenesis. A previous report revealed that betatrophin mRNA is induced by the thyroid hormone in HepG2 cells. Subsequent studies confirmed that transcriptional regulation is dependent on the thyroid hormone receptor that binds to the betatrophin upstream element. Therefore, betatrophin is a novel gene dramatically activated by the thyroid hormone. However, there is no evidence to date showing that TH is capable of regulating betatrophin expression in human beings. The current study investigated the change of betatrophin levels in patients with hyperthyroidism before and after thionamide treatment and explored the association of serum betatrophin levels with hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hyperthyroidism
* Must be drug-naive before recruitment

Exclusion Criteria:

* diabetes
* hypertension
* cancer
* pregnancy
* lactation
* subacute thyroiditis
* postpartum thyroiditis
* abnormal liver function
* abnormal kidney function
* infectious diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with hyperthyroidism would be recruited from the Department of Endocrinology, the First People's Hospital of Xuzhou, from May, 2016, to May, 2017. During the same period, the healthy controls would be selected.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Serum betatrophin levels | Change from baseline at 3 months

SECONDARY OUTCOMES:
Thyroid function index | At baseline and at the end of the third month
blood lipid profile | At baseline and at the end of the third month
liver function index | At baseline and at the end of the third month
hypersensitive c-reactive protein (hs-CRP) | At baseline and at the end of the third month
Blood glucose | At baseline and at the end of the third month
Serum insulin levels | At baseline and at the end of the third month

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhaoling, BD, Study Chair — The First People's Hospital of Xuzhou; Hu Hao, MD, Study Director — The First People's Hospital of Xuzhou; Gao Zhaohua, MD, Principal Investigator — The First People's Hospital of Xuzhou; Zhou Tingting, MD, Principal Investigator — The First People's Hospital of Xuzhou; Yin Wenwen, MD, Principal Investigator — The First People's Hospital of Xuzhou; Cai Ruonan, MD, Principal Investigator — The First People's Hospital of Xuzhou
Locations (1):
- The First People's Hospital of Xuzhou,, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators are committed to the open and timely dissemination of the research outcomes. Plans for sharing resources with the scientific community include presentations and publications in peer-reviewed journals. The final data set will be made available to the public upon completion of the study.

REFERENCES:
- [Background] Lopez D, Abisambra Socarras JF, Bedi M, Ness GC. Activation of the hepatic LDL receptor promoter by thyroid hormone. Biochim Biophys Acta. 2007 Sep;1771(9):1216-25. doi: 10.1016/j.bbalip.2007.05.001. Epub 2007 May 21. PMID 17572141
- [Background] Ribeiro MO, Carvalho SD, Schultz JJ, Chiellini G, Scanlan TS, Bianco AC, Brent GA. Thyroid hormone--sympathetic interaction and adaptive thermogenesis are thyroid hormone receptor isoform--specific. J Clin Invest. 2001 Jul;108(1):97-105. doi: 10.1172/JCI12584. PMID 11435461
- [Background] Dong XY, Pang XW, Yu ST, Su YR, Wang HC, Yin YH, Wang YD, Chen WF. Identification of genes differentially expressed in human hepatocellular carcinoma by a modified suppression subtractive hybridization method. Int J Cancer. 2004 Nov 1;112(2):239-48. doi: 10.1002/ijc.20363. PMID 15352036
- [Background] Quagliarini F, Wang Y, Kozlitina J, Grishin NV, Hyde R, Boerwinkle E, Valenzuela DM, Murphy AJ, Cohen JC, Hobbs HH. Atypical angiopoietin-like protein that regulates ANGPTL3. Proc Natl Acad Sci U S A. 2012 Nov 27;109(48):19751-6. doi: 10.1073/pnas.1217552109. Epub 2012 Nov 12. PMID 23150577
- [Background] Ren G, Kim JY, Smas CM. Identification of RIFL, a novel adipocyte-enriched insulin target gene with a role in lipid metabolism. Am J Physiol Endocrinol Metab. 2012 Aug 1;303(3):E334-51. doi: 10.1152/ajpendo.00084.2012. Epub 2012 May 8. PMID 22569073
- [Background] Zhang R. Lipasin, a novel nutritionally-regulated liver-enriched factor that regulates serum triglyceride levels. Biochem Biophys Res Commun. 2012 Aug 10;424(4):786-92. doi: 10.1016/j.bbrc.2012.07.038. Epub 2012 Jul 15. PMID 22809513
- [Background] Yi P, Park JS, Melton DA. Betatrophin: a hormone that controls pancreatic beta cell proliferation. Cell. 2013 May 9;153(4):747-58. doi: 10.1016/j.cell.2013.04.008. Epub 2013 Apr 25. PMID 23623304 (Retraction: PMID 28038792 Cell. 2017 Jan 12;168(1-2):326)
- [Result] Tseng YH, Ke PY, Liao CJ, Wu SM, Chi HC, Tsai CY, Chen CY, Lin YH, Lin KH. Chromosome 19 open reading frame 80 is upregulated by thyroid hormone and modulates autophagy and lipid metabolism. Autophagy. 2014 Jan;10(1):20-31. doi: 10.4161/auto.26126. Epub 2013 Nov 11. PMID 24262987
- See also: test link — http://www.ncbi.nlm.nih.gov/pubmed
- Available data/document: Individual Participant Data Set — https://www.opendrive.com/ — Using network platform: https://www.opendrive.com/ username: 18361811955@163.com password: woaini1314 The repository and management of the data can be obtained via "Public Folder".